CLINICAL TRIAL: NCT02697058
Title: Phase II Randomized Study of BAX2398 in Combination With 5-Fluorouracil and Calcium Levofolinate in Japanese Patients With Metastatic Pancreatic Cancer, Which Progressed or Recurred After Prior Gemcitabine-Based Therapy
Brief Title: Phase II of BAX2398/5-FU/Calcium Levofolinate in Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 331501
Record Dates: First submitted 2016-02-20; First posted 2016-03-03 (Estimated); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — irinotecan sucrosofate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: Yes

ARMS (3):
- Part 1: Safety and PK (Experimental): BAX2398 in combination with 5-FU/calcium levofolinate
  Interventions: Biological: BAX2398 + 5-FU/calcium levofolinate
- Part 2: Safety, PK, Efficacy (Experimental): BAX2398 in combination with 5-FU/calcium levofolinate
  Interventions: Biological: BAX2398 + 5-FU/calcium levofolinate
- Part 2: 5-FU/calcium levofolinate alone (Active Comparator): 5-FU/calcium levofolinate
  Interventions: Drug: 5-FU/calcium levofolinate

INTERVENTIONS:
Biological: BAX2398 + 5-FU/calcium levofolinate — BAX2398 (a liposomal formulation of irinotecan) in combination with 5-FU/calcium levofolinate
  Other Names: nal-IRI; MM-398
  Arms: Part 1: Safety and PK; Part 2: Safety, PK, Efficacy
Drug: 5-FU/calcium levofolinate — 5-FU/calcium levofolinate alone
  Arms: Part 2: 5-FU/calcium levofolinate alone

SUMMARY:
Study Part 1: To assess the safety and tolerability, and to characterize the pharmacokinetics (PK) of BAX2398 in combination with 5-FU/calcium levofolinate in Japanese patients.

Study Part 2: To compare the efficacy of BAX2398 in combination with 5-FU/calcium levofolinate versus 5-FU/calcium levofolinate as assessed by Progression Free Survival (PFS) using Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1).

ELIGIBILITY:
Inclusion Criteria:

1. Participant is ≥20 years of age at the time of screening.
2. Histologically or cytologically confirmed adenocarcinoma of exocrine pancreas
3. Documented metastatic disease
4. Metastatic disease with at least one measurable lesion as defined by RECIST 1.1 guidelines
5. Documented disease progression after prior gemcitabine or any gemcitabine containing therapy but excluding irinotecan, for locally advanced or metastatic setting. Prior chemotherapy must be stopped for at least 21 days before the first dose.
6. Karnofsky Performance Status (KPS) ≥70
7. Adequate bone marrow reserves
8. Adequate hepatic function
9. Adequate renal function
10. Normal ECG including Fridericia corrected QT interval (QTcF) <440 ms within 7 days prior to first dose of study drug
11. Recovered from the effects of any prior surgery, radiotherapy or other anti-neoplastic therapy with no residual adverse events (AEs) of Grade ≥2.
12. Able to understand and sign an informed consent (or have a legal representative who is able to do so)
13. If female of childbearing potential, participant presents with a negative pregnancy, and agrees to employ adequate birth control measures during the study dosing period and for 3 months following the last dose of study drug.
14. Participant is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

1. Active and uncontrolled central nervous system (CNS) metastases; for controlled CNS metastases, patient should have been off steroids for at least 28 days prior to starting study therapy.
2. History of any second malignancy in the last 5 years; participants with prior history of in-situ cancer or basal or squamous cell skin cancers are eligible. Participants with other malignancies are eligible if they have been continuously disease free for at least 5 years.
3. Severe arterial thromboembolic events (myocardial infarction, unstable angina pectoris, stroke) less than 6 months before inclusion.
4. Cannot stop medications that are potent CYP3A4 inducers within 2 weeks and inhibitors within 1 week before start of treatment.
5. Significant cardiac conduction abnormalities, including a history of long QTcF syndrome and/or pacemaker.
6. New York Heart Association (NYHA) Class III or IV congestive heart failure, ventricular arrhythmias or uncontrolled blood pressure.
7. Active infection, including active hepatitis B virus (HBV), hepatitis C virus (HCV), and HIV, or an unexplained fever >38.5°C during screening visits or on the first scheduled day of dosing (at the discretion of the investigator, patients with tumor fever may be enrolled), which in the investigator's opinion might compromise the patient's participation in the trial or affect the study outcome.
8. Known hypersensitivity to any of the components of BAX2398, other liposomal products, fluoropyrimidines, or calcium levofolinate.
9. Any other medical or social condition deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.
10. Participant has been exposed to an investigational product (IP) within 30 days prior to the first dose of the study drug or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study.
11. Participant is a family member or employee of the investigator.
12. Participant is pregnant or lactating at the time of enrollment. Lactating mothers can resume breast feeding 30 days following the last dose of the study treatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) in Part 2 of Study | Part 2 Baseline to the end of the study (up to 22 months)
  Progression Free Survival (PFS) was defined as the time from randomization to the first documented disease progression based on the independent central review board's assessment using RECIST 1.1 or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) in Part 1 of Study | Part 1 Baseline to the end of the study (up to 22 months)
  Progression Free Survival (PFS) was defined as the time from randomization to the first documented disease progression based on the independent central review board's assessment using RECIST 1.1 or death due to any cause, whichever occurred first.
Overall Survival (OS) | Baseline to the end of the study (up to 22 months)
  OS was defined as the time from the date of informed consent (Part 1) or date of randomization (Part 2) to death due to any cause or the date of last known alive.
Time to Treatment Failure (TTF) | Baseline to the end of the study (up to 22 months)
  TTF was defined as the time from randomization to disease progression according to RECIST 1.1, death due to any cause, discontinuation of treatment due to toxicity, or for symptomatic deterioration, or start of another anticancer therapy
Objective Response Rate (ORR) | Baseline to the end of the study (up to 22 months)
  ORR was defined as the proportion of participants with a best overall response of complete response (CR) or partial response (PR)
Disease Control Rate (DCR) | Baseline to the end of the study (up to 22 months)
  DCR was defined as the proportion of participants with a best overall response of complete response (CR); partial response (PR); or stable disease (SD) lasting >=24 weeks
Tumor Marker Response | Baseline, every 6 weeks and 37 days post last visit (up to 22 months)
  Tumor marker response was defined as decrease of 50% of cancer antigen (CA)-19-9 in relation to the baseline level at least once during the treatment period. Tumor marker response evaluable population consist of participants who have elevated CA-19-9 level (greater than [<] 30 international unit [IU] / millilitre [ml]) at baseline and at least one post baseline CA-19-9 assessment.
Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Scores | Baseline, Day 1 of Cycle 4, 7, 10, 13, and 16; and 37 days post last visit (up to 22 months)
  The EORTC-QLQC30 is a reliable and valid measure of the quality of life of cancer participants in multicultural clinical research settings. It incorporates nine multi-item scales: five functional scales (physical [PFS], role [RFS], cognitive [CFS], emotional [EFS], and social [SFS]); three symptom scales (fatigue [FSS], pain [PSS], and nausea and vomiting [NVSS]); and a global health status (GHS) and quality-of-life scale. Several single-item symptom measures are also included. All scales and single-item measures range=0 to 100. High score for a functional scale=high/healthy level of functioning. High score for global health status/QoL=high QoL. High score for symptom scale/single item=high level of symptomatology/problems.
Change From Baseline in Pain | Baseline, Days 1 and 8 of Cycles 1, 2, 4, 5, 7, 8, 10, 11, 13, 14, 16, 17, Day 1 of Cycles 3, 6, 9, 12, 15, 18 and 37 days post last visit (up to 22 months)
  Participants assessed pain on the VAS. VAS range: 0 (no pain) to 100 worst pain.
Change from Baseline in Analgesic use | Baseline, Days 1 and 8 of Cycles 1, 2, 4, 5, 7, 8, 10, 11, 13, 14, 16, 17, Day 1 of Cycles 3, 6, 9, 12, 15, 18 and 37 days post last visit (up to 22 months)
  Participants recorded their analgesic usage in diaries.
Number of Participants With Karnofsky Performance Score (KPS) | Baseline, Day 1 of Cycles 1 - 18 and 37 days post last visit (up to 22 months)
  The Karnofsky score runs from 100 to 0, where 100 is "perfect" health and 0 is death.
Change From Baseline in Weight | Baseline, Days 1 and 8 of Cycles 1, 2, 4, 5, 7, 8, 10, 11, 13, 14, 16, 17, Day 1 of Cycles 3, 6, 9, 12, 15, 18 and 37 days post last visit (up to 22 months)
  The participant defined to be a clinical benefit responder if the weight change is classified as Positive. (1) Positive: an increase of at least 7% over baseline, maintained for at least 2 cycles (2) Non-positive: any other change in weight.
Number of Participants With Serious Adverse Events | From start of study treatment up to 22 months
  A Serious adverse event (AE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Number of Participants With Non-Serious Adverse Events | From start of study treatment up to 22 months
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment.
Number of Participants With Clinically Significant Findings From the Physical Examination | From start of study treatment up to 22 months
  Physical examination done on the following body systems: general appearance, head and neck, eyes and ears, nose and throat, chest, lungs, heart, abdomen, extremities and joints, lymph nodes, skin, and neurological.
Number of Participants With Clinically Significant Changes in Vital Signs | From start of study treatment up to 22 months
  Number of participants with clinically significant changes in vital signs assessed by measuring height, weight, temperature, respiration rate, pulse rate, systolic and diastolic blood pressure, and body surface area at all the listed time points was reported.
Number of Participants With Clinically Significant Changes in Laboratory Results | From start of study treatment up to 22 months
  Number of participants with clinically significant changes in laboratory results was reported.
Number of Participants With Clinically Significant Changes in Twelve-lead Electrocardiogram (ECG) | From start of study treatment up to 22 months
  Number of participants with clinically significant changes in ECG results was reported.
Maximum Plasma Concentration (Cmax) of Total Irinotecan in Study Part 1 | Cycle 1: pre dose, 30, 60, 90 minutes after start of infusion and 1, 3, 9, 24, 36, 48, 72, 120 and 168 hours after the end of the infusion; Cycle 2: pre dose
  The Cmax of total irinotecan (encapsulated + unencapsulated) in study part 1 was reported.
Maximum Plasma Concentration (Cmax) of Total Primary Metabolite of Irinotecan (SN-38) in Study Part 1 | Cycle 1: pre dose, 30, 60, 90 minutes after start of infusion and 1, 3, 9, 24, 36, 48, 72, 120 and 168 hours after the end of the infusion; Cycle 2: pre dose
  The Cmax of total SN-38 (encapsulated + unencapsulated) in study part 1 was reported.
Maximum Plasma Concentration (Cmax) of SN-38-Glucuronide (SN-38G) in Study Part 1 | Cycle 1: pre dose, 30, 60, 90 minutes after start of infusion and 1, 3, 9, 24, 36, 48, 72, 120 and 168 hours after the end of the infusion; Cycle 2: pre dose
  The Cmax of SN-38G in study part 1 was reported.
Time of Maximum Concentration (tmax) of Total Irinotecan, Total SN-38, and SN-38-Glucuronide (SN-38G) in Study Part 1 | Cycle 1: pre dose, 30, 60, 90 minutes after start of infusion and 1, 3, 9, 24, 36, 48, 72, 120 and 168 hours after the end of the infusion; Cycle 2: pre dose
  The Tmax of total irinotecan (encapsulated + unencapsulated), total SN-38 (encapsulated + unencapsulated), and SN-38G was reported.
Terminal Half-Life (t1/2) of Total Irinotecan, Total SN-38, and SN-38-Glucuronide (SN-38G) in Study Part 1 | Cycle 1: pre dose, 30, 60, 90 minutes after start of infusion and 1, 3, 9, 24, 36, 48, 72, 120 and 168 hours after the end of the infusion; Cycle 2: pre dose
  The t1/2 of Total irinotecan (encapsulated + unencapsulated), total SN-38 (encapsulated + unencapsulated), and SN-38-glucuronide (SN-38G) in study part 1 was reported.
Area Under the Concentration-time Curve in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-infinity) of Total Irinotecan in Study Part 1 | Cycle 1: pre dose, 30, 60, 90 minutes after start of infusion and 1, 3, 9, 24, 36, 48, 72, 120 and 168 hours after the end of the infusion; Cycle 2: pre dose
  The AUC0-infinity of Total irinotecan (encapsulated + unencapsulated) in study part 1 was reported.
Area Under the Concentration-time Curve in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-infinity) of Total SN-38 in Study Part 1. | Cycle 1: pre dose, 30, 60, 90 minutes after start of infusion and 1, 3, 9, 24, 36, 48, 72, 120 and 168 hours after the end of the infusion; Cycle 2: pre dose
  The AUC0-infinity of total SN-38 (encapsulated + unencapsulated)in study part 1 was reported.
Area Under the Concentration-time Curve in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-infinity) of SN-38-Glucuronide (SN-38G) IN Study Part 1. | Cycle 1: pre dose, 30, 60, 90 minutes after start of infusion and 1, 3, 9, 24, 36, 48, 72, 120 and 168 hours after the end of the infusion; Cycle 2: pre dose
  The AUC0-infinity of SN-38-glucuronide (SN-38G) in study part 1 was reported.
Systemic Clearance (CL) of Total Irinotecan in Study Part 1 | Cycle 1: pre dose, 30, 60, 90 minutes after start of infusion and 1, 3, 9, 24, 36, 48, 72, 120 and 168 hours after the end of the infusion; Cycle 2: pre dose
  The CL of total irinotecan (encapsulated + unencapsulated) in study part 1 was reported.
Systemic Clearance (CL) of Total SN-38 in Study Part 1 | Cycle 1: pre dose, 30, 60, 90 minutes after start of infusion and 1, 3, 9, 24, 36, 48, 72, 120 and 168 hours after the end of the infusion; Cycle 2: pre dose
  The CL of SN-38 (encapsulated + unencapsulated), in study part 1 was reported.
Systemic Clearance (CL) of SN-38-Glucuronide (SN-38G) in Study Part 1 | Cycle 1: pre dose, 30, 60, 90 minutes after start of infusion and 1, 3, 9, 24, 36, 48, 72, 120 and 168 hours after the end of the infusion; Cycle 2: pre dose
  The CL of SN-38-glucuronide (SN-38G) in study part 1 was reported.
Volume of Distribution (V) of Total Irinotecan in Study Part 1 | Cycle 1: pre dose, 30, 60, 90 minutes after start of infusion and 1, 3, 9, 24, 36, 48, 72, 120 and 168 hours after the end of the infusion; Cycle 2: pre dose
  The V of total irinotecan (encapsulated + unencapsulated) in study part 1 was reported.
Volume of Distribution (V) of Total SN-38 in Study Part 1. | Cycle 1: pre dose, 30, 60, 90 minutes after start of infusion and 1, 3, 9, 24, 36, 48, 72, 120 and 168 hours after the end of the infusion; Cycle 2: pre dose
  The V of total SN-38 (encapsulated + unencapsulated), in study part 1 was reported.
Volume of Distribution (V) of SN-38-Glucuronide (SN-38G) in Study Part 1. | Cycle 1: pre dose, 30, 60, 90 minutes after start of infusion and 1, 3, 9, 24, 36, 48, 72, 120 and 168 hours after the end of the infusion; Cycle 2: pre dose
  The V of SN-38-glucuronide (SN-38G) in study part 1 was reported.
Volume of Distribution at Steady-State (Vss) of Total Irinotecan in Study Part 1 | Cycle 1: pre dose, 30, 60, 90 minutes after start of infusion and 1, 3, 9, 24, 36, 48, 72, 120 and 168 hours after the end of the infusion; Cycle 2: pre dose
  The Vss of total irinotecan (encapsulated + unencapsulated) in study part 1 was reported.
Volume of Distribution at Steady-state (Vss) of Total SN-38 in Study Part 1 | Cycle 1: pre dose, 30, 60, 90 minutes after start of infusion and 1, 3, 9, 24, 36, 48, 72, 120 and 168 hours after the end of the infusion; Cycle 2: pre dose
  The Vss of total irinotecan (encapsulated + unencapsulated), SN-38 (encapsulated + unencapsulated), and SN-38-glucuronide (SN-38G) was reported.
Volume of Distribution at Steady-state (Vss) of SN-38-Glucuronide (SN-38G) in Study Part 1 | Cycle 1: pre dose, 30, 60, 90 minutes after start of infusion and 1, 3, 9, 24, 36, 48, 72, 120 and 168 hours after the end of the infusion; Cycle 2: pre dose
  The Vss of SN-38-glucuronide (SN-38G) in study part 1 was reported.
Terminal Half-life (t1/2) - Total Irinotecan, SN-38, and SN-38-Glucuronide (SN-38G) | Cycle 1: pre dose, 15-90 minutes after start of infusion; and 0-6, 6-24, 24-48, 72-168, and 216-264 hours after the end of the infusion; Cycle 2: pre dose
  The t1/2 of total irinotecan (encapsulated + unencapsulated), SN-38 (encapsulated + unencapsulated), and SN-38-glucuronide (SN-38G) was reported.
Area Under the Curve (AUC) - Total Irinotecan, SN-38, and SN-38-Glucuronide (SN-38G) | Cycle 1: pre dose, 15-90 minutes after start of infusion; and 0-6, 6-24, 24-48, 72-168, and 216-264 hours after the end of the infusion; Cycle 2: pre dose
  The AUC of total irinotecan (encapsulated + unencapsulated), SN-38 (encapsulated + unencapsulated), and SN-38-glucuronide (SN-38G) was reported.
Systemic Clearance (CL) -Total Irinotecan, SN-38, and SN-38-Glucuronide (SN-38G) | Cycle 1: pre dose, 15-90 minutes after start of infusion; and 0-6, 6-24, 24-48, 72-168, and 216-264 hours after the end of the infusion; Cycle 2: pre dose
  The CL of total irinotecan (encapsulated + unencapsulated), SN-38 (encapsulated + unencapsulated), and SN-38-glucuronide (SN-38G) was reported.
Volume of Distribution (V)-Total Irinotecan, SN-38, and SN-38-Glucuronide (SN-38G) | Cycle 1: pre dose, 15-90 minutes after start of infusion; and 0-6, 6-24, 24-48, 72-168, and 216-264 hours after the end of the infusion; Cycle 2: pre dose
  The V of total irinotecan (encapsulated + unencapsulated), SN-38 (encapsulated + unencapsulated), and SN-38-glucuronide (SN-38G) was reported.
Volume of Distribution at Steady-State (Vss)-Total Irinotecan, SN-38, and SN-38-Glucuronide (SN-38G) | Cycle 1: pre dose, 15-90 minutes after start of infusion; and 0-6, 6-24, 24-48, 72-168, and 216-264 hours after the end of the infusion; Cycle 2: pre dose
  The Vss of total irinotecan (encapsulated + unencapsulated), SN-38 (encapsulated + unencapsulated), and SN-38-glucuronide (SN-38G) was reported.

CONTACTS AND LOCATIONS:
Locations (16):
- Japan (16):
  - Hirosaki University School of Medicine & Hospital, Hirosaki-shi, Aomori
  - Chiba Cancer Center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - NHO Shikoku Cancer Center, Matsuyama, Ehime
  - NHO Kyushu Cancer Center, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa -ku
  - Kyoto University Hospital, Kyoto, Kyoto
  - NHO Osaka National Hospital, Osaka, Osaka
  - Osaka International Cancer Institute, Osaka, Osaka
  - Saitama Cancer Center, Kitaadachi-gun, Saitama
  - National Cancer Center Hospital, Chuo Ku, Tokyo
  - Cancer Institute Hospital of JFCR, Kōtoku, Tokyo-To
  - Kyorin University Hospital, Mitaka-shi, Tokyo-To

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  They can ask for all interventional clinical studies:
  * submitted for new medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier or an affiliate are the Marketing Authorization Holders (MAH). The date of the first Marketing Authorization of the new medicine (or the new indication) in one of the EEA Member States will be considered within this scope.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- [Background] Ueno M, Nakamori S, Sugimori K, Kanai M, Ikeda M, Ozaka M, Furukawa M, Okusaka T, Kawabe K, Furuse J, Komatsu Y, Ishii H, Sato A, Shimizu S, Chugh P, Tang R, Ioka T. nal-IRI+5-FU/LV versus 5-FU/LV in post-gemcitabine metastatic pancreatic cancer: Randomized phase 2 trial in Japanese patients. Cancer Med. 2020 Dec;9(24):9396-9408. doi: 10.1002/cam4.3558. Epub 2020 Oct 25. PMID 33099898
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: study-level clinical trial data — https://clinicaltrials.servier.com/